CLINICAL TRIAL: NCT00248248
Title: A Phase II Non-randomized Study of DOXIL Consolidation Treatment for Ovarian Cancer, Cancer of the Fallopian Tube or Peritoneal Carcinoma.
Brief Title: DOXIL for Consolidation Therapy in Ovarian Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southeastern Gynecologic Oncology (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEGO_DOXIL_CONS2005
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Ovarian Neoplasm
Keywords: Consolidation; Ovarian cancer; DOXIL; Hand-foot syndrome
MeSH Terms: conditions — Ovarian Neoplasms; Hand-Foot Syndrome | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: liposomal doxorubicin — Doxil at 50mg/m2 infused over one hour every 3 or 4 weeks for 3-6 cycles

SUMMARY:
The primary objective for this study is to evaluate the development, frequency and severity of hand foot syndrome (HFS) in ovarian cancer subjects treated with Doxil®, as consolidation therapy, on an every two week schedule.

The secondary objective for this study is to assess one-year progression free survival rate (PFS).

DETAILED DESCRIPTION:
While the majority of subjects with advanced ovarian cancer will respond well to the initial chemotherapy regimen of taxol/platinum, these responses are generally of limited duration. Even women who have a surgically defined complete response to initial chemotherapy have >50% recurrence rate in Stage III disease. Once ovarian cancer has recurred it is rare that cure is possible, therefore, there is a critical need to define new therapeutic strategies in the treatment of ovarian cancer. Consolidation chemotherapy is one possible strategy. The strategy behind consolidation chemotherapy institutes second-line chemotherapy immediately following a clinical response but before evidence of recurrence. This strategy has gained popularity with many oncologists, secondary to the results of GOG 178, a large study by the Southwest Oncology Group and the Gynecologic Oncology Group. GOG 178 set out to explore both efficacy and patient tolerability in the consolidation setting. Moreover, the objective of the GOG 178 study was to compare two different durations of consolidation treatment using taxol consolidation in clinically NED ovarian cancer subjects following primary chemotherapy of carbo/taxol. The results of GOG178 suggested that a longer course (12 vs. 3 cycles of paclitaxel) gave subjects a longer median progression-free survival (28 vs. 21 months). This trial was closed early due to a statistically improved PFS in subjects receiving 12-month regimen of paclitaxel versus the 3 month regimen. Unfortunately, we will never definitively learn if this improved PFS translates to improved survival for ovarian cancer patients. A limitation of this regimen is the cumulative and sometimes irreversible side effect of neuropathy. Doxil has been selected in this consolidation trial due to documented success in second- line setting with ovarian cancer subjects without long term negative sequelae such as neuropathy The anthracycline antibiotic doxorubicin has a broad spectrum of antineoplastic action and a correspondingly widespread degree of clinical use. In addition to its role in the treatment of ovarian cancer, doxorubicin is indicated in the treatment of Hodgkin's disease and non-Hodgkin's lymphoma, hepatocellular and gastric carcinoma, small cell cancer of the lung, soft tissue and bone sarcomas, as well as cancer of the breast, bladder, and thyroid. Unfortunately, toxicity limits the therapeutic activity of doxorubicin and may preclude adequate dosing.

The conventional formulation of the drug is rapidly cleared from the bloodstream and has a very large volume of distribution, which may contribute to the drug's toxicity. High cumulative doses of doxorubicin generally must be avoided because of the potential for cardiotoxicity, while individual doses are often limited by myelosuppression. Alopecia typically develops and persists throughout treatment. Severe acute nausea and vomiting, stomatitis, and esophagitis are additional adverse effects of doxorubicin that may necessitate dose-reduction or discontinuation of the drug. A doxorubicin formulation with improved tolerability might increase the drug's therapeutic ratio and thus enhance its efficacy.

Liposomal encapsulation of doxorubicin may reduce both the nonspecific drug delivery to normal tissues as well as the high peak plasma levels of free drug responsible for its toxicity. At the same time, a liposomal formulation may deliver doxorubicin to tumors with improved specificity. Doxil is a doxorubicin formulation in which the drug is encapsulated in liposomes (Stealthâ liposomes) that escape instant recognition and uptake by the mononuclear phagocyte system. As a result, the formulation has a long circulation time, and the liposomes can eventually become extravasated through the abnormally permeable vessels characteristic of many tumors. Once concentrated in tumors the liposomes of Doxil can deliver high levels of doxorubicin to malignant cells, without affecting normal tissue.1

Doxil is approved by the FDA for use in subjects with ovarian cancer whose disease has progressed or recurred after platinum-based chemotherapy and in subjects with HIV Kaposi's Sarcoma. Doxil established efficacy as a single agent in recurrent ovarian cancer as a result of three open-label, single-arm clinical studies of 176 subjects with metastatic ovarian cancer. Subjects in these studies received Doxil at 50mg/m2 infused over one hour every 3 or 4 weeks for 3-6 cycles or longer in the absence of dose-limiting toxicity or progression of disease. Doxil has been used for several years as a 2nd line chemotherapy agent. In the randomized Phase III study of subjects with recurrent ovarian cancer by Gordon et al, there was an 18% reduction in the risk of death for subjects treated with Doxil (median survival 62.7weeks) compared to topotecan (median survival 59.7 weeks). In platinum sensitive subjects (who recurred after more than six months), the reduction in risk of death was even more dramatic, a 30% reduction was noted in the subjects who received Doxil (median survival 107.9 weeks) versus topotecan (median survival 70.1 weeks). In this trial Doxil 50mg/m2 was administered every 28 days, resulting in 23.4% of the subjects with grade 3 or 4 hand foot syndrome (HFS). 4 Management of this side effect included increasing the dosage interval and/or decreasing the dose by 25%. Today, Doxil 40mg/m2 every 28 days is commonly used for treatment of recurrent ovarian cancer. Rose et al reported their results from a retrospective review noting the 40mg/m2 dose every 28 days minimizes toxicity without sacrificing efficacy.6

Experience has taught us this toxicity can be minimized with patient education focusing on alteration of activities in the day preceding and 3-5 days follow drug administration. Other side effects such as bone marrow suppression, alopecia, nausea, vomiting, and fatigue are minimal. There have been several small trials using weekly and bi-weekly Doxil® in cancer patients, including breast, gastric, pancreatic and colon cancer, in an attempt to reduce the incidence of hand foot syndrome with encouraging results

This study will evaluate the efficacy of Doxil in clinically NED ovarian cancer subjects following standard platinum/taxane based therapy. Applying every two-week dosing of Doxil 20mg/m2 as this is expected to minimize the most problematic side effect, HFS.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a initial histopathologic diagnosis of epithelial ovarian cancer, cancer of the fallopian tube or primary peritoneal carcinoma
2. Subjects must have completed front-line platinum based chemotherapy with or without a taxane and be clinically NED (CA 125 <35, negative CT scan, normal physical exam).
3. Subjects must not have had other chemotherapy, radiation, hormonal, or biotherapy within four weeks of initiating Doxil therapy.
4. Doxil treatment must begin within 6 weeks following last cycle of initial chemotherapy.
5. Subjects may have a second look laparoscopy, however, there must be no gross disease present (microscopic disease or pathologically negative).
6. Subjects must have adequate renal function: creatinine < 2.5 mg/dL (< 200 mmol/L).
7. Subjects must have adequate liver functions: total bilirubin </=1.5 x upper limit of normal (ULN), transaminases (AST/ALT) </=2.5 x ULN
8. Subjects must have adequate bone marrow function: Platelets >100,000 cells/mm3, Hemoglobin > 9.0g/dL and ANC > 1,500 cells/mm3.
9. Subjects must be age 18 or greater.
10. Subjects must have signed approved informed consent.
11. Subjects must have a Zubrod Performance Status of 0 or 1. (Appendix A)
12. With the exception of non-melanoma skin cancer, subjects with other invasive malignancies who had (or have) any evidence of the other cancer present within the last 5 years, or whose previous cancer treatment contraindicates this protocol therapy are excluded.
13. Subjects must have no other major systemic medical illness expected to affect survival.
14. Subjects with a life expectancy > 12 weeks.
15. Subjects must have a MUGA scan or 2-d echocardiogram indicating an ejection fraction (LVEF) of > than 50% within 42 days prior to first dose of study drug. The method used at baseline must be used for final monitoring.

Exclusion Criteria:

1. Prior therapy with Doxil, anthracyclines, or anthracendedione. History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin HCL or the components of Doxil®
2. Prior radiation therapy to more than one-third of the hematopoietic sites.
3. Myocardial infarct within 6 months before enrollment, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities. See Appendix B (New York State Heart Association Classification).
4. Uncontrolled systemic infection or history of any other unstable serious condition or illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2005-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Development, frequency, and severity of hand-foot syndrome with every two week therapy | 5 years

SECONDARY OUTCOMES:
One-year progression free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Hines, MD, FACOG, Principal Investigator — Southeastern Gynecologic Oncology
Locations (1):
- Southeastern Gynecologic Oncology, Atlanta, Georgia, United States

REFERENCES:
- [Background] Gordon AN, Tonda M, Sun S, Rackoff W; Doxil Study 30-49 Investigators. Long-term survival advantage for women treated with pegylated liposomal doxorubicin compared with topotecan in a phase 3 randomized study of recurrent and refractory epithelial ovarian cancer. Gynecol Oncol. 2004 Oct;95(1):1-8. doi: 10.1016/j.ygyno.2004.07.011. PMID 15385103
- [Background] Rose PG, Maxson JH, Fusco N, Mossbruger K, Rodriguez M. Liposomal doxorubicin in ovarian, peritoneal, and tubal carcinoma: a retrospective comparative study of single-agent dosages. Gynecol Oncol. 2001 Aug;82(2):323-8. doi: 10.1006/gyno.2001.6272. PMID 11531287